CLINICAL TRIAL: NCT04032171
Title: A Phase III, Multicenter, Randomized, Parallel Group, Double Blind, Double Dummy, Active Controlled Study of Evobrutinib Compared With an Interferon Beta 1a (Avonex®), in Participants With RMS to Evaluate Efficacy and Safety
Brief Title: Study of Evobrutinib in Participants With RMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following analysis of open label extension (OLE) data from RMS phase 2 study (MS200527- 0086), it was determined that a change in active comparator warranted in phase 3 RMS comprised of trial MS200527-0074. Consequently, this trial terminated early.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200527_0074; 2018-004700-19 (EudraCT Number)
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Evobrutinib; Avonex®; Interferon-beta 1a; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — evobrutinib; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evobrutinib + Avonex® matched Placebo (Experimental): Participants received active evobrutinib twice daily (BID) along with concomitant intramuscular (IM) injection of placebo matched to Avonex® once a week. Treatment period was planned to be of 96 weeks.
  Interventions: Drug: Evobrutinib; Drug: Avonex® matched Placebo
- Avonex® + Evobrutinib matched Placebo (Active Comparator): Participants received IM injection of active Avonex® once a week along with concomitant placebo matched to evobrutinib BID. Treatment period was planned to be of 96 weeks.
  Interventions: Drug: Avonex®; Drug: Evobrutinib matched Placebo

INTERVENTIONS:
Drug: Evobrutinib — Participants received evobrutinib twice daily (BID).
  Other Names: M2951
  Arms: Evobrutinib + Avonex® matched Placebo
Drug: Avonex® — Participants received avonex® IM injection once a week.
  Arms: Avonex® + Evobrutinib matched Placebo
Drug: Avonex® matched Placebo — Participants received IM injection of placebo matched to avonex® once a week.
  Arms: Evobrutinib + Avonex® matched Placebo
Drug: Evobrutinib matched Placebo — Participants received placebo matched to evobrutinib twice a day.
  Arms: Avonex® + Evobrutinib matched Placebo

SUMMARY:
The study was to evaluate the efficacy and safety of evobrutinib administered orally twice daily versus Interferon-beta-1a (Avonex®), once a week intramuscularly in participants with Relapsing Multiple Sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with RMS (relapsing-remitting multiple sclerosis [RRMS] or secondary progressive multiple sclerosis [SPMS] with relapses) in accordance with 2017 Revised McDonald criteria (Thompson 2018).
* Participants with one or more documented relapses within the 2 years before Screening with either: a. one relapse which occurred within the last year prior to randomization, OR b. the presence of at least 1 gadolinium-enhancing (Gd+) T1 lesion within 6 months prior to randomization.
* Participants have EDSS score of 0 to 5.5 at Baseline. Participants with an EDSS score <= 2 at screening are only eligible for participation if their disease duration (time since onset of symptoms) is no more than 10 years.
* Participants are neurologically stable for >= 30 days prior to both screening and baseline.
* Female participants must be neither pregnant nor breast-feeding and must lack child-bearing potential, as defined by either: post-menopausal or surgically sterile or use an effective method of contraception for the duration of the study.
* Participants have given written informed consent prior to any study-related procedure.
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants diagnosed with Progressive MS, in accordance with the 2017 Revised McDonald criteria as follows: a). Participants with Primary Progressive MS. b). Participants with secondary progressive MS without evidence of relapse.
* Disease duration more than (>) 10 years in participants with an EDSS =< 2.0 at screening.
* Immunologic disorder other than MS, or any other condition requiring oral, intravenous (IV) , intramuscular, or intra-articular corticosteroid therapy, with the exception of well-controlled Type 2 diabetes mellitus or well controlled thyroid disease.
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (2):
- Please Contact U.S. Medical Information, Rockland, Massachusetts, United States
- Please Contact the Communication Center, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html.

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0074
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was to be conducted in 2 periods; double blind period and open label extension period. However, due to early termination of the study, the sponsor decided not to conduct the open label extension period. A total of 950 participants were planned to be included in 1:1 to treatment with evobrutinib or Avonex, however only 1 participant was enrolled in evobrutinib due to early termination.
Period: Overall Study
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Study Termination | 1 | 0

BASELINE CHARACTERISTICS:
Population: Following analysis of open label extension (OLE) data from RMS phase 2 study (MS200527- 0086), it was determined that a change in active comparator warranted in phase 3 RMS comprised of trial MS200527-0074. Consequently, this trial terminated early, therefore no participants enrolled in Avonex® + Evobrutinib matched Placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: The annualized relapse rate at 96 weeks was to be calculated based on qualified relapses. A qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to MS. The relapse should be accompanied by an increase of 0.5 points or more on Expanded Disability Status Scale (EDSS), or 2 points increase on one of the Functional System Scores (FSS), or 1 point increase on at least two of the FSS. The increase in FSS scores must be related to the neurological symptoms which were reported as new or worsening.
Time Frame: At Week 96
Population: Following analysis of open label extension (OLE) data from RMS phase 2 study (MS200527- 0086), it was determined that a change in active comparator warranted in phase 3 RMS comprised of trial MS200527-0074. Consequently, this trial terminated early, therefore, it was decided as per Statistical Analysis Plan not to report the efficacy data for this study.
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to First Occurrence of 12-Week Confirmed Expanded Disability Status Scale (EDSS) Progression
Description: EDSS is an ordinal scale in half-point increments that measures disability in participants with MS. EDSS progression is defined as an increase of 1 point or more from Baseline EDSS score when the Baseline score is 5.0 or less, and an increase of 0.5 points or more when the Baseline score is 5.5 or greater. Time to first occurrence of 12-week confirmed EDSS progression is defined as the time from randomization to the first EDSS progression event that was confirmed at a regularly scheduled visit at least 12 weeks later.
Time Frame: Baseline up to 96 weeks
Population: as for outcome 1
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to First Occurrence of 24-Week Confirmed Expanded Disability Status Scale (EDSS) Progression
Description: EDSS is an ordinal scale in half-point increments that measures disability in participants with MS. EDSS progression is defined as an increase of 1 point or more from Baseline EDSS score when the Baseline score is 5.0 or less, and an increase of 0.5 points or more when the Baseline score is 5.5 or greater. Time to first occurrence of 24-week confirmed EDSS progression is defined as the time from randomization to the first EDSS progression event that was confirmed at a regularly scheduled visit at least 24 weeks later.
Time Frame: Baseline up to 96 weeks
Population: as for outcome 1
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Short Form Score at Week 96
Description: The PROMIS PF Short Form is specific to measuring the physical function domain of MS patients, with each item on the form scored on a T-score metric. Higher scores indicate higher PF. Change from baseline at Week 96 is the difference between the PROMIS PF scores at 96 weeks and at baseline.
Time Frame: Baseline, Week 96
Population: as for outcome 1
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form Score at Week 96
Description: The PROMIS Fatigue Short Form is specific to measuring the fatigue domain of MS patients, with each item on the form scored on a T-score metric. Higher scores indicate higher fatigue. Change from baseline at Week 96 is the difference between the PROMIS Fatigue scores at 96 weeks and at baseline.
Time Frame: Baseline, Week 96
Population: as for outcome 1
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Total Number of Gadolinium-Enhancing (Gd+) Time Constant 1 (T1) Lesions Assessed by Magnetic Resonance Imaging (MRI) Scans at Week 24, 48, and 96
Description: Total number of Gd+ T1 lesions was to be assessed using magnetic resonance imaging (MRI).
Time Frame: At Week 24, 48 and 96
Population: as for outcome 1
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Total Number of New or Enlarging Time Constant 2 (T2) Lesions Assessed by Magnetic Resonance Imaging (MRI) Scans at Week 24, 48, and 96
Description: Total number of new or enlarging T2 lesions was to be assessed using magnetic resonance imaging (MRI).
Time Frame: At Week 24, 48 and 96
Population: as for outcome 1
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, regardless if it is considered related to the medicinal product. TEAE is an AE that started after study drug treatment; or if the event was continuous from baseline & was serious, related to investigational medicinal product (IMP), or resulted in death, discontinuation, interruption or reduction of study therapy. TEAEs included both serious and non-serious TEAEs. AESIs included liver AEs (possible drug-induced, non-infectious, non-alcoholic and immune-mediated) infections (serious and opportunistic infections), lipase and amylase elevation, and seizure.
Time Frame: Baseline up to 254 days
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Participants
  Participants with AESIs | 0 |
  Participants with TEAEs | 1 |
  Participants with Serious TEAEs | 0 |

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on Severity According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in participant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs included both serious TEAEs and non-serious TEAEs. Severity of TEAEs were graded using NCI CTCAE v4.03 toxicity grades, as follows: Grade 1= Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with TEAEs based on severity were reported.
Time Frame: Baseline up to 254 days
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Participants
  Grade 1 | 1 |
  Grade 2 | 0 |
  Grade 3 | 0 |
  Grade 4 | 0 |
  Grade 5 | 0 |

10. Secondary Outcome: Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time points.
Time Frame: At Day 1, Week 2 unscheduled 1, Week 12 and Early Discontinuation (ED) (up to approximately 36 weeks
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: Millimeters of mercury (mmHg)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Millimeters of mercury (mmHg)
  DBP: Day 1 | 72 |
  DBP: Week 2 unscheduled 1 | 68 |
  DBP: Week 12 | 76 |
  DBP: ED (up to approximately 36 weeks) | 84 |
  SBP: Day 1 | 124 |
  SBP: Week 2 unscheduled 1 | 119 |
  SBP: Week 12 | 130 |
  SBP:ED (up to approximately 36 weeks) | 140 |

11. Secondary Outcome: Vital Signs: Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points.
Time Frame: At Day 1, Week 2 unscheduled 1, Week 12 and Early Discontinuation ED (up to approximately 36 weeks)
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: Beats per minute
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Beats per minute
  Pulse rate: Day 1 | 71 |
  Pulse rate: Week 2 unscheduled 1 | 77 |
  Pulse rate: Week 12 | 75 |
  Pulse rate: ED (up to approximately 36 weeks) | 80 |

12. Secondary Outcome: Vital Signs: Respiratory Rate
Description: Respiration rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points.
Time Frame: At Day 1, Week 2 unscheduled 1, Week 12 and Early Discontinuation ED (up to approximately 36 weeks)
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: Breaths Per Minute
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Breaths Per Minute
  Respiratory rate: Day 1 | 12 |
  Respiratory rate: Week 2 unscheduled 1 | 18 |
  Respiratory rate: Week 12 | 12 |
  Respiratory rate: ED (up to approximately 36 weeks) | 14 |

13. Secondary Outcome: Vital Signs: Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest for the participants at indicated time points.
Time Frame: At Day 1, Week 2 unscheduled 1, Week 12 and Early Discontinuation (ED) (up to approximately 36 weeks)
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: Degree celsius
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Degree celsius
  Day 1 | 36.4 |
  Week 2 unscheduled 1 | 36.7 |
  Week 12 | 36.9 |
  ED (up to approximately 36 weeks) | 36.7 |

14. Secondary Outcome: Vital Signs: Weight
Time Frame: At Day 1, Week 2 unscheduled 1, Week 12 and Early Discontinuation (up to approximately 36 weeks)
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: kilogram (kg)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
kilogram (kg)
  Day 1 | 91.4 |
  Week 2 unscheduled 1 | 92.3 |
  Week 12 | 92.6 |
  ED (up to approximately 36 weeks) | 95.5 |

15. Secondary Outcome: Number of Participants With Abnormal Lab Values
Description: The total number of participants with laboratory test abnormalities was assessed. Clinical laboratory tests included hematology, coagulation, biochemistry and urinalysis.
Time Frame: Baseline up to 254 days
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Participants | 0 |

16. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: ECG parameters included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals.
Time Frame: Baseline up to 254 days
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
Participants | 0 |

17. Secondary Outcome: Absolute Concentrations of Immunoglobulin (Ig) A Level
Description: Absolute concentrations of Immunoglobulin (Ig) A was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: gram per liter (g/L)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
gram per liter (g/L)
  Day 1 | 0.8 |
  Day 92 | 0.92 |

18. Secondary Outcome: Absolute Concentrations of Immunoglobulin (Ig) G Level
Description: Absolute concentrations of Immunoglobulin (Ig) E was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: grams per liter (g/L)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
grams per liter (g/L)
  Day 1 | 5.54 |
  Day 92 | 6.11 |

19. Secondary Outcome: Absolute Concentrations of Immunoglobulin (Ig) M Level
Description: Absolute concentrations of Immunoglobulin (Ig) M was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: grams per liter (g/L)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
grams per liter (g/L)
  Day 1 | 0.29 |
  Day 92 | 0.25 |

20. Secondary Outcome: Absolute Concentrations of Immunoglobulin (Ig) E Level
Description: Absolute concentrations of Immunoglobulin (Ig) E was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: International units per milliliter
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
International units per milliliter
  Day 1 | 14.1 |
  Day 92 | 16.7 |

21. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) A Level
Description: Change from baseline in immunoglobulin (Ig) A level was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: gram per liter (g/L)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
gram per liter (g/L) | 0.12 |

22. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) E Level
Description: Change from baseline in immunoglobulin (Ig) E level was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: International units per milliliter
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
International units per milliliter | 2.6 |

23. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) G Level
Description: Change from baseline in immunoglobulin (Ig) G level was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: grams per liter (g/L)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
grams per liter (g/L) | 0.57 |

24. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) M Level
Description: Change from baseline in immunoglobulin (Ig) M level was reported.
Time Frame: At Day 1 and Day 92
Population: SAF analysis set included all participants who were administered any dose of any study intervention.
Measure: Number; unit: grams per liter (g/L)
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
Number analyzed (Participants) | 1 | 0
grams per liter (g/L) | -0.04 |

ADVERSE EVENTS:
Time Frame: Baseline up to 254 days
Description: Following analysis of open label extension (OLE) data from RMS phase 2 study (MS200527- 0086), it was determined that a change in active comparator warranted in phase 3 RMS comprised of trial MS200527-0074. Consequently, this trial terminated early, therefore no participants enrolled in Avonex® + Evobrutinib matched Placebo arm.
Arm/Group | Evobrutinib + Avonex® Matched Placebo | Avonex® + Evobrutinib Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evobrutinib + Avonex® Matched Placebo (N=1) | Avonex® + Evobrutinib Matched Placebo (N=0)
Dry eye (Eye disorders) | 1 | 0
Peripheral edema (Nervous system disorders) | 1 | 0
Hypercholesterolemia (Hepatobiliary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Following analysis of open label extension (OLE) data from RMS phase 2 study (MS200527- 0086), it was determined that a change in active comparator warranted in phase 3 RMS comprised of trial MS200527-0074. Consequently, this trial terminated early, therefore, it was decided as per Statistical Analysis Plan not to report the efficacy data for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04032171/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT04032171/SAP_001.pdf